CLINICAL TRIAL: NCT01160211
Title: A Phase III Trial to Compare the Safety and Efficacy of Lapatinib Plus Trastuzumab Plus an Aromatase Inhibitor (AI) vs. Trastuzumab Plus an AI vs. Lapatinib Plus an AI as 1st- or 2nd- Line Therapy in Postmenopausal Subjects With Hormone Receptor+, HER2-positive Metastatic Breast Cancer (MBC) Who Received Prior Trastuzumab and Endocrine Therapies
Brief Title: A Study to Compare the Safety and Efficacy of an Aromatase Inhibitor in Combination With Lapatinib, Trastuzumab or Both for the Treatment of Hormone Receptor Positive, HER2+ Metastatic Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 114299; 2010-019577-16 (EudraCT Number); CLAP016A2307 (Other: Novartis)
Record Dates: First submitted 2010-07-01; First posted 2010-07-12 (Estimated); Results first posted 2019-07-15 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Neoplasms, Breast
Keywords: 1st line MBC; MBC; hormone receptor positive; lapatinib; trastuzumab; HER2 positive; aromatase inhibitor
MeSH Terms: conditions — Breast Neoplasms | interventions — Lapatinib; Trastuzumab; Aromatase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment group A (Experimental): Lapatinib 1000 mg PO once daily + Trastuzumab (loading dose of 8 mg/kg) followed by the maintenance dose of 6 mg/kg IV every 3 weeks (q3weeks) + an Aromatase Inhibitor (AI) of Investigator's choice PO once daily.
  Interventions: Drug: Lapatinib; Drug: Trastuzumab; Drug: Aromatase Inhibitor
- Treatment group B (Active Comparator): Trastuzumab (loading dose of 8 mg/kg) followed by maintenance dose of 6 mg/kg IV every 3 weeks (q3weeks) + an Aromatase Inhibitor (AI) of Investigator's choice PO once daily.
  Interventions: Drug: Trastuzumab; Drug: Aromatase Inhibitor
- Treatment Group C (Active Comparator): Lapatinib 1500 mg PO once daily + an Aromatase Inhibitor (AI) of Investigator's choice PO once daily.
  Interventions: Drug: Aromatase Inhibitor; Drug: Lapatinib

INTERVENTIONS:
Drug: Lapatinib — 1000 mg by mouth once a day
  Arms: Treatment group A
Drug: Trastuzumab — Loading dose of 8 mg/kg IV followed by the maintenance dose of 6 mg/kg IV every 3 weeks (q3weeks)
  Arms: Treatment group A; Treatment group B
Drug: Aromatase Inhibitor — Aromatase inhibitor (either letrozole, anastrozole, or exemestane) of investigator's choice given by mouth once daily
Drug: Lapatinib — 1500 mg by mouth once daily
  Arms: Treatment Group C

SUMMARY:
A study to compare the safety and efficacy of an aromatase inhibitor in combination with lapatinib, trastuzumab or both for the treatment of hormone receptor positive, HER2+ metastatic breast cancer (MBC).

DETAILED DESCRIPTION:
This Phase III, multicenter, open-label study randomized subjects to one of the three treatment arms:

1. Treatment group A: lapatinib 1000 mg PO once daily + trastuzumab (loading dose of 8 mg/kg) followed by the maintenance dose of 6 mg/kg IV q3weeks + an AI (either letrozole, anastrozole, or exemestane) of Investigator's choice PO once daily.
2. Treatment group B: trastuzumab (loading dose of 8 mg/kg) followed by maintenance dose of 6 mg/kg IV q3weeks + an AI (either letrozole, anastrozole, or exemestane) of Investigator's choice PO once daily.
3. Treatment group C: lapatinib 1500 mg PO once daily + an AI (either letrozole, anastrozole, or exemestane) of Investigator's choice PO once daily.

Treatment continued until disease progression, death, or unacceptable toxicities, whichever came first.

Subjects who discontinued study treatment for reasons other than disease progression were followed-up every 12 weeks until disease progression or death, until the start of post-study treatment anti-cancer therapy (including radiotherapy and surgery), withdrawal of consent, or lost to follow-up, whichever came first.

ELIGIBILITY:
Inclusion Criteria

Subjects eligible for enrollment in the study must meet all of the following criteria:

1. Signed written informed consent. In Korea and Japan, subjects between >=18 and <20 years of age must also have a legal representative sign the written informed consent.
2. Post-menopausal female subjects >=18 years of age. Post-menopausal as defined by any of the following:

   * Subjects at least 60 years of age.
   * Subjects under 60 years of age and amenorrhic for at least 12 consecutive months AND follicle-stimulating hormone (FSH) and estradiol levels in postmenopausal range (utilizing ranges from the local laboratory facility).
   * Prior bilateral oophorectomy.
   * Prior radiation castration with amenorrhea for at least 6 months
3. Subjects must have a history of histologically confirmed breast cancer, with a clinically confirmed diagnosis of metastatic disease [confirmed by histology, cytology or other clinical means (e.g. CT, MRI)]. Subjects may have either measurable or non-measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST 1.1)
4. Tumors that are ER+ and/or PgR+ by local laboratory
5. Documentation of HER2 overexpression or gene amplification, in the invasive component of either the primary tumor or metastatic disease site as defined as:

   * 3+ by Immunohistochemistry (IHC) and/or
   * HER2/neu gene amplification by fluorescence, chromogenic or silver in situ hybridization [FISH, CISH or SISH; >6 HER2/neu gene copies per nucleus or a FISH, CISH or SISH test ratio (HER2 gene copies to chromosome 17 signals) of ≥2.0]
6. Subject must have received at least one prior regimen containing trastuzumab in combination with chemotherapy for breast cancer:.

   * Subject has ONLY received prior trastuzumab in combination with chemotherapy as neoadjuvant and/or adjuvant treatment. OR
   * Subject has received ONE prior trastuzumab-containing regimen for metastatic disease (and has progressed), and may or may not have received prior trastuzumab in combination with chemotherapy as neoadjuvant and/or adjuvant treatment.
7. Subject must have received prior endocrine therapy (such as aromatase inhibitors or selective estrogen receptor modulators). 8. Subjects who have a life expectancy of > 6 months as assessed by the treating investigator

9. Subjects must have baseline Left Ventricular Ejection Fraction (LVEF) ≥50% measured by echocardiography (ECHO) or multi-gated acquisition scan (MUGA) 10. Subject must have an ECOG performance status of 0-1 11. All prior treatment related toxicities must be CTCAE (Version 4.0) ≤ Grade 1 at the time of randomization 12. Completion of screening assessments 13. Adequate baseline organ function. 14. Subjects must meet all of the following criteria:

* QTc <450msec or
* QTc <480msec for subjects with bundle branch block The QTc is the QT interval corrected for heart rate according to either Bazett's formula (QTcB) or to Fridericia's formula (QTcF), machine or manual over read, for males and females. The specific formula that will be used in a protocol should be determined prior to initiation of the study, and the formula used to determine inclusion and discontinuation should be the same throughout the study. The QTc should be based on single or averaged QTc values of triplicate electrocardiograms (ECGs) obtained over a brief recording period

Exclusion criteria:

1. History of another malignancy. Exception: Subjects who have been disease-free for 5 years, or subjects with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible.
2. Subjects with extensive symptomatic visceral disease including hepatic involvement and pulmonary lymphangitic spread of tumor, or the disease is considered by the investigator to be rapidly progressing or life threatening (subjects who are intended for chemotherapy)
3. Serious cardiac illness or medical condition including but not confined to:

   * Uncontrolled arrhythmias
   * Uncontrolled or symptomatic angina
   * History of congestive heart failure (CHF)
   * Documented myocardial infarction <6 months from study entry
4. Known history of, or clinical evidence of, central nervous system (CNS) metastases or leptomeningeal carcinomatosis
5. Have acute or currently active/requiring anti-viral therapy hepatic or biliary disease (with the exception of subjects with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment)
6. Have a concurrent disease or condition that may interfere with study participation, or any serious medical disorder that would interfere with the subject's safety (for example, active or uncontrolled infection or any psychiatric condition prohibiting understanding or rendering of informed consent)
7. Have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels
8. Have a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to any of the study agents or their excipients that, in the opinion of the Investigator or GSK medical monitor, contraindicates their participation
9. Any prohibited medication.
10. Administration of an investigational drug within 30 days or 5 half-lives, whichever is longer, preceding the first dose of study treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 369 (Actual)
Dates: Start 2011-05-05 (Actual); Primary Completion 2016-03-11 (Actual); Study Completion 2022-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (101):
- United States (4):
  - Novartis Investigative Site, Hollywood, Florida
  - Novartis Investigative Site, Augusta, Georgia
  - Novartis Investigative Site, Germantown, Tennessee
  - Novartis Investigative Site, Tacoma, Washington
- Argentina (10):
  - Novartis Investigative Site, Berazategui, Buenos Aires
  - Novartis Investigative Site, Capital Federal, Buenos Aires
  - Novartis Investigative Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Novartis Investigative Site, La Plata, Buenos Aires
  - Novartis Investigative Site, Viedma, Río Negro Province
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, La Rioja
  - Novartis Investigative Site, Quilmes
  - Novartis Investigative Site, San Miguel de Tucumán
- Australia (2):
  - Novartis Investigative Site, Albury
  - Novartis Investigative Site, Douglas
- Belgium (2):
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Namur
- Brazil (5):
  - Novartis Investigative Site, Goiânia, Goiás
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Barretos, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
  - Novartis Investigative Site, Rio de Janeiro
- Bulgaria (3):
  - Novartis Investigative Site, Plovdiv
  - Novartis Investigative Site, Sofia
  - Novartis Investigative Site, Varna
- China (5):
  - Novartis Investigative Site, Fuzhou, Fujian
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Changchun, Jilin
  - Novartis Investigative Site, Harbin
  - Novartis Investigative Site, Shanghai
- Croatia (2):
  - Novartis Investigative Site, Osijek
  - Novartis Investigative Site, Zagreb
- France (3):
  - Novartis Investigative Site, Besançon
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Paris
- Germany (5):
  - Novartis Investigative Site, Munich, Bavaria
  - Novartis Investigative Site, Fürstenwalde, Brandenburg
  - Novartis Investigative Site, Goslar, Lower Saxony
  - Novartis Investigative Site, Troisdorf, North Rhine-Westphalia
  - Novartis Investigative Site, Velbert, North Rhine-Westphalia
- Greece (3):
  - Novartis Investigative Site, Alexandroupoli
  - Novartis Investigative Site, Chania
  - Novartis Investigative Site, Heraklion
- Hong Kong (3):
  - Novartis Investigative Site, Hong Kong
  - Novartis Investigative Site, Kowloon
  - Novartis Investigative Site, Tuenmen
- Hungary (8):
  - Novartis Investigative Site, Győr
  - Novartis Investigative Site, Gyula
  - Novartis Investigative Site, Kaposvár
  - Novartis Investigative Site, Miskolc
  - Novartis Investigative Site, Nyíregyháza
  - Novartis Investigative Site, Pécs
  - Novartis Investigative Site, Szeged
  - Novartis Investigative Site, Zalaegerszeg
- India (2):
  - Novartis Investigative Site, Nagpur
  - Novartis Investigative Site, New Delhi
- Israel (3):
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Ramat Gan
- Novartis Investigative Site, Rozzano (MI), Lombardy, Italy
- Japan (6):
  - Novartis Investigative Site, Aichi
  - Novartis Investigative Site, Chiba
  - Novartis Investigative Site, Ehime
  - Novartis Investigative Site, Osaka
  - Novartis Investigative Site, Saitama
  - Novartis Investigative Site, Tokyo
- Peru (2):
  - Novartis Investigative Site, Arequipa
  - Novartis Investigative Site, Lima
- Poland (2):
  - Novartis Investigative Site, Konin
  - Novartis Investigative Site, Warsaw
- Portugal (2):
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Porto
- Russia (5):
  - Novartis Investigative Site, Arkhangelsk
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Ryazan
  - Novartis Investigative Site, Saint Petersburg
- Serbia (2):
  - Novartis Investigative Site, Belgrade
  - Novartis Investigative Site, Kamenitz
- Novartis Investigative Site, Singapore, Singapore
- South Korea (2):
  - Novartis Investigative Site, Gyeonggi-do
  - Novartis Investigative Site, Seoul
- Spain (4):
  - Novartis Investigative Site, A Coruña
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Castellon
  - Novartis Investigative Site, Madrid
- Taiwan (3):
  - Novartis Investigative Site, Changhua
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Taipei
- Turkey (Türkiye) (2):
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Izmir
- Ukraine (6):
  - Novartis Investigative Site, Chernivtsi
  - Novartis Investigative Site, Kharkiv
  - Novartis Investigative Site, Liutizh
  - Novartis Investigative Site, Sumy
  - Novartis Investigative Site, Uzhhorod
  - Novartis Investigative Site, Vinnitsia
- United Kingdom (3):
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Maidstone
  - Novartis Investigative Site, Peterborough

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Background] Johnston SRD, Hegg R, Im SA, Park IH, Burdaeva O, Kurteva G, Press MF, Tjulandin S, Iwata H, Simon SD, Kenny S, Sarp S, Izquierdo MA, Williams LS, Gradishar WJ. Phase III, Randomized Study of Dual Human Epidermal Growth Factor Receptor 2 (HER2) Blockade With Lapatinib Plus Trastuzumab in Combination With an Aromatase Inhibitor in Postmenopausal Women With HER2-Positive, Hormone Receptor-Positive Metastatic Breast Cancer: ALTERNATIVE. J Clin Oncol. 2018 Mar 10;36(8):741-748. doi: 10.1200/JCO.2017.74.7824. Epub 2017 Dec 15. PMID 29244528 (Retraction: PMID 32822279 J Clin Oncol. 2021 Jan 1;39(1):95)
- [Derived] Johnston SRD, Hegg R, Im SA, Park IH, Burdaeva O, Kurteva G, Press MF, Tjulandin S, Iwata H, Simon SD, Kenny S, Sarp S, Izquierdo MA, Williams LS, Gradishar WJ. Phase III, Randomized Study of Dual Human Epidermal Growth Factor Receptor 2 (HER2) Blockade With Lapatinib Plus Trastuzumab in Combination With an Aromatase Inhibitor in Postmenopausal Women With HER2-Positive, Hormone Receptor-Positive Metastatic Breast Cancer: Updated Results of ALTERNATIVE. J Clin Oncol. 2021 Jan 1;39(1):79-89. doi: 10.1200/JCO.20.01894. Epub 2020 Aug 21. PMID 32822287

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 113 centers in 29 countries worldwide (Argentina, Australia, Belgium, Brazil, Bulgaria, China, Croatia, France, Germany, Greece, Hong Kong, Hungary, India, Israel, Italy, Japan, Peru, Poland, Portugal, Republic of Korea, Russia, Serbia, Singapore, Spain, Taiwan, Turkey, UK, Ukraine and USA)
Groups:
- Lapatinib + Trastuzumab + Aromatase Inhibitor (AI): Lapatinib 1000 mg PO once daily + Trastuzumab (loading dose of 8 mg/kg) followed by the maintenance dose of 6 mg/kg IV every 3 weeks (q3weeks) + an Aromatase Inhibitor (AI) of Investigator's choice PO once daily.
- Lapatinib + Aromatase Inhibitor (AI): Lapatinib 1500 mg PO once daily + an Aromatase Inhibitor (AI) of Investigator's choice PO once daily.
- Trastuzumab + Aromatase Inhibitor (AI): Trastuzumab (loading dose of 8 mg/kg) followed by maintenance dose of 6 mg/kg IV every 3 weeks (q3weeks) + an Aromatase Inhibitor (AI) of Investigator's choice PO once daily.
Period: Overall Study
Arm/Group | Lapatinib + Trastuzumab + Aromatase Inhibitor (AI) | Lapatinib + Aromatase Inhibitor (AI) | Trastuzumab + Aromatase Inhibitor (AI)
Started (All randomized subjects regardless of whether or not treatment was administered (Intent-to-Treat (ITT) Set)) | 124 | 123 | 122
Safety Set (All randomized subjects who received at least one dose of study treatment and was based on the actual treatment received if this differed from that to which the subject was randomized) | 123 | 123 | 121
Completed | 64 | 64 | 55
Not Completed | 60 | 59 | 67
Not completed — Subject Reached Protocol-Defined Stopping Criteria | 49 | 49 | 59
Not completed — Lost to Follow-up | 4 | 8 | 4
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 2 | 2
Not completed — Data unavailable due to regulatory issues | 2 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lapatinib + Trastuzumab + Aromatase Inhibitor (AI) | Lapatinib + Aromatase Inhibitor (AI) | Trastuzumab + Aromatase Inhibitor (AI) | Total
Number analyzed (Participants) | 124 | 123 | 122 | 369
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.9 (11.15) | 57.1 (9.98) | 54.9 (10.10) | 56.3 (10.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 124 | 123 | 122 | 369
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 1 | 3
  Asian | 31 | 31 | 32 | 94
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 4 | 3 | 10
  White | 89 | 85 | 84 | 258
  More than one race | 0 | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) Events in Lapatinib + Trastuzumab + Aromatase Inhibitor (AI) vs. Trastuzumab + Aromatase Inhibitor (AI)
Description: The Number of Participants with Progression free survival (PFS) events in the Lapatinib + Trastuzumab + Aromatase Inhibitor (AI) arm vs. Trastuzumab + Aromatase Inhibitor (AI) arm was based on assessments by the Investigator.
Time Frame: From date of randomization until date of progression or date of death from any cause, whichever comes first, assessed up approximately 5 years
Population: Participants in the Intent-to-Treat (ITT) Population with available data for the outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Lapatinib + Trastuzumab + Aromatase Inhibitor (AI) | Trastuzumab + Aromatase Inhibitor (AI)
Number analyzed (Participants) | 120 | 117
Participants
  Disease progression or died (event) | 62 | 75
  Censored, follow-up for disease progression ended | 7 | 3
  Censored, f/p for disease progression ongoing | 51 | 39
Statistical Analysis 1: Comparison: Lapatinib + Trastuzumab + Aromatase Inhibitor (AI) vs Trastuzumab + Aromatase Inhibitor (AI); Null hypothesis H0: λ ≥ 1 or to reject it in favor of the alternative hypothesis HA: λ <1, where λ is the hazard ratio (HR) between Treatment Group A and Treatment Group B for progression-free survival; Test type: Superiority; p = 0.0063, Log Rank — Pike estimate of the treatment hazard ratio, <1 indicates a lower risk compared with trastuzumab + AI; using a two-sided stratified log-rank test (based on stratification factors); Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.45 to 0.88]

2. Primary Outcome: Median Kaplan Meier Estimates for PFS in Lapatinib + Trastuzumab + Aromatase Inhibitor (AI) vs. Trastuzumab + Aromatase Inhibitor (AI)
Description: Progression free survival (PFS) was defined as the interval of time between the date of randomization and the earliest date of disease progression (with radiological evidence) or death from any cause, or to the date of censor. Disease progression was based on assessments by the Investigator.
Time Frame: as for outcome 1
Population: Participants in the Intent-to-Treat (ITT) Population with available data for the outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lapatinib + Trastuzumab + Aromatase Inhibitor (AI) | Trastuzumab + Aromatase Inhibitor (AI)
Number analyzed (Participants) | 120 | 117
Months | 11.0 [8.3 to 13.8] | 5.6 [5.4 to 8.3]

3. Secondary Outcome: Progression Free Survival (PFS)
Description: as for outcome 2
Time Frame: From date of randomization until date of progression or date of death from any cause, whichever comes first, assessed up approximately 11 years
Population: Intent-to-Treat (ITT) Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lapatinib + Trastuzumab + Aromatase Inhibitor (AI) | Lapatinib + Aromatase Inhibitor (AI) | Trastuzumab + Aromatase Inhibitor (AI)
Number analyzed (Participants) | 124 | 123 | 122
Months | 11.1 [10.0 to 15.3] | 8.3 [7.1 to 11.0] | 5.7 [5.5 to 8.3]
Statistical Analysis 1: Comparison: Lapatinib + Trastuzumab + Aromatase Inhibitor (AI) vs Trastuzumab + Aromatase Inhibitor (AI); Test type: Superiority; Hazard Ratio (HR) = 0.59, 95% CI 2-sided [0.44 to 0.79]
Statistical Analysis 2: Comparison: Lapatinib + Aromatase Inhibitor (AI) vs Trastuzumab + Aromatase Inhibitor (AI); Test type: Superiority; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.66 to 1.15]
Statistical Analysis 3: Comparison: Lapatinib + Trastuzumab + Aromatase Inhibitor (AI) vs Lapatinib + Aromatase Inhibitor (AI); Test type: Superiority; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.51 to 0.92]

4. Secondary Outcome: Overall Survival (OS)
Description: The Number of Participants with Overall Survival (OS) events was based on assessments by the Investigator.
Time Frame: From date of randomization until date of death from any cause, assessed up approximately 11 years
Population: Intent-to-Treat (ITT) Population
Measure: Count of Participants; unit: Participants
Arm/Group | Lapatinib + Trastuzumab + Aromatase Inhibitor (AI) | Lapatinib + Aromatase Inhibitor (AI) | Trastuzumab + Aromatase Inhibitor (AI)
Number analyzed (Participants) | 124 | 123 | 122
Participants
  Death | 38 | 45 | 39
  Censored, follow-up ended | 86 | 78 | 83
  Censored, follow-up ongoing | 0 | 0 | 0

5. Secondary Outcome: Overall Response Rate (ORR)
Description: Overall Response Rate (ORR) was defined as the proportion of participants achieving either a Complete Response (CR) or Partial Response (PR). The ORR was calculated from the Investigator's assessment of response based on RECIST 1.1. Subjects with an unknown or missing response were treated as non-responders; i.e. they were included in the denominator when calculating the percentages. Subjects who do not have measurable disease contributed to the Response Rate based analyses, for the evaluation of CR, SD and PD.
Time Frame: Up approximately 11 years
Population: Intent-to-Treat (ITT) Population.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Lapatinib + Trastuzumab + Aromatase Inhibitor (AI) | Lapatinib + Aromatase Inhibitor (AI) | Trastuzumab + Aromatase Inhibitor (AI)
Number analyzed (Participants) | 124 | 123 | 122
Percentage of Participants | 32.3 [24.2 to 41.2] | 22.8 [15.7 to 31.2] | 17.2 [11.0 to 25.1]

6. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: Clinical Benefit Rate (CBR) was defined as the percentage of patients with evidence of Complete Response (CR), Partial Response (PR), or maintaining Stable Disease (SD) for at least 6 months while on study, according to the investigator assessment of response per RECIST 1.1 criteria.
Time Frame: Up approximately 11 years
Population: Intent-to-Treat (ITT) Population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Lapatinib + Trastuzumab + Aromatase Inhibitor (AI) | Lapatinib + Aromatase Inhibitor (AI) | Trastuzumab + Aromatase Inhibitor (AI)
Number analyzed (Participants) | 124 | 123 | 122
Percentage of Participants | 51.6 [42.5 to 60.7] | 43.1 [34.2 to 52.3] | 34.4 [26.1 to 43.6]

7. Secondary Outcome: Time to Response
Description: Time to Response (TTR) was defined as the time from randomization to the earliest date of Complete Response (CR) or Partial Response (PR)
Time Frame: From date of randomization until the earliest date of Complete Response (CR) or Partial Response (PR), assessed up approximately 11 years
Population: Intent-to-Treat (ITT) Population. Only participants achieving either a confirmed complete response (CR) or partial response (PR)
Measure: Median (Full Range); unit: Days
Arm/Group | Lapatinib + Trastuzumab + Aromatase Inhibitor (AI) | Lapatinib + Aromatase Inhibitor (AI) | Trastuzumab + Aromatase Inhibitor (AI)
Number analyzed (Participants) | 40 | 28 | 21
Days | 85.0 [72 to 1031] | 86.5 [65 to 1175] | 86.0 [67 to 337]

8. Secondary Outcome: Duration of Response (DoR)
Description: Duration of Response (DOR) was defined as the duration between the date of first documented Complete Response (CR) or Partial Response (PR) and the date of first documented sign of Progressive Disease or Death, or to the date of censor.
Time Frame: From first documented evidence of CR or PR (the response prior to confirmation) until time of documented disease progression or death due to any cause, whichever comes first, assessed up approximately 11 years
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lapatinib + Trastuzumab + Aromatase Inhibitor (AI) | Lapatinib + Aromatase Inhibitor (AI) | Trastuzumab + Aromatase Inhibitor (AI)
Number analyzed (Participants) | 40 | 28 | 21
Months | 22.5 [11.1 to 33.1] | 11.1 [5.6 to NA] — Not estimable due to insufficient number of participants with events | 11.8 [5.4 to 28.1]

9. Secondary Outcome: Mean Change in the Quality of Life (QoL) Status Relative to Baseline FACT-B Overall and Subscale Scores at Last On Treatment Assessment
Description: Quality of life was assessed using the Functional Assessment of Cancer Therapy-Breast (FACT-B) questionnaire. It is a 37-item (27 general questions and 10 breast cancer specific questions) self-reporting instrument consisting of 5 dimensions: physical well-being (PWB), social well-being (SWB), emotional well-being (EWB), functional well-being (FWB), and a breast cancer subscale (BCS). The followings were the score ranges for each self-reporting subscale: • PWB : 0-28 • SWB : 0-28 • EWB : 0-24 • FWB : 0-28 • BCS : 0-40 FACT-B Total Outcome Index (TOI) = PWB + FWB + BCS (range:0 - 96) FACT-B Total Score = PWB + SWB + EWB + FWB + BCS (range:0-148) FACT-G Total Score = PWB + SWB + EWB + FWB (range:0-108). For all the FACIT scales and symptom indices, the higher the score the better QoL
Time Frame: Day 1 (pre-dose), up approximately 11 years
Population: Participants in the Intent-to-Treat (ITT) Population with available data for the outcome measure.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Lapatinib + Trastuzumab + Aromatase Inhibitor (AI) | Lapatinib + Aromatase Inhibitor (AI) | Trastuzumab + Aromatase Inhibitor (AI)
Number analyzed (Participants) | 115 | 113 | 110
score on a scale
  FACT-B total score: number analyzed (Participants) | 114 | 110 | 110
  FACT-B total score | -4.2 (1.48) | -6.3 (1.51) | -2.4 (1.51)
  FACT-G total score: number analyzed (Participants) | 114 | 111 | 110
  FACT-G total score | -4.3 (1.22) | -5.9 (1.24) | -2.8 (1.24)
  FACT-B trial outcome Index (TOI): number analyzed (Participants) | 114 | 111 | 110
  FACT-B trial outcome Index (TOI) | -3.3 (1.05) | -4.2 (1.07) | -0.6 (1.07)
  Physical well-being (PWB) | -2.0 (0.48) | -2.1 (0.49) | -0.5 (0.49)
  Social family wellbeing (SWB): number analyzed (Participants) | 115 | 112 | 110
  Social family wellbeing (SWB) | -0.5 (0.50) | -1.5 (0.50) | -0.9 (0.51)
  Emotional wellbeing (EWB) | -0.4 (0.40) | -0.6 (0.40) | -1.0 (0.41)
  Functional wellbeing (FWB) | -1.3 (0.45) | -1.7 (0.46) | -0.3 (0.46)
  Breast cancer subscale (BCS) | 0.0 (0.47) | -0.5 (0.47) | 0.4 (0.48)
Statistical Analysis 1: Comparison: Lapatinib + Trastuzumab + Aromatase Inhibitor (AI) vs Trastuzumab + Aromatase Inhibitor (AI); FACT-B total score; Test type: Superiority; Least square difference = -1.79, 95% CI 2-sided [-5.95 to 2.36], Standard Error of Mean 2.111
Statistical Analysis 2: Comparison: Lapatinib + Aromatase Inhibitor (AI) vs Trastuzumab + Aromatase Inhibitor (AI); FACT-B total score; Test type: Superiority; Least square difference = -3.90, 95% CI 2-sided [-8.09 to 0.29], Standard Error of Mean 2.130
Statistical Analysis 3: Comparison: Lapatinib + Trastuzumab + Aromatase Inhibitor (AI) vs Trastuzumab + Aromatase Inhibitor (AI); FACT-G total score; Test type: Superiority; Least square difference = -1.50, 95% CI 2-sided [-4.92 to 1.92], Standard Error of Mean 1.739
Statistical Analysis 4: Comparison: Lapatinib + Aromatase Inhibitor (AI) vs Trastuzumab + Aromatase Inhibitor (AI); FACT-G total score; Test type: Superiority; Least square difference = -3.10, 95% CI 2-sided [-6.55 to 0.34], Standard Error of Mean 1.751
Statistical Analysis 5: Comparison: Lapatinib + Trastuzumab + Aromatase Inhibitor (AI) vs Trastuzumab + Aromatase Inhibitor (AI); FACT-B trial outcome index (TOI); Test type: Superiority; Least square difference = -2.70, 95% CI 2-sided [-5.66 to 0.25], Standard Error of Mean 1.502
Statistical Analysis 6: Comparison: Lapatinib + Aromatase Inhibitor (AI) vs Trastuzumab + Aromatase Inhibitor (AI); FACT-B trial outcome index (TOI); Test type: Superiority; Least square difference = -3.61, 95% CI 2-sided [-6.59 to -0.64], Standard Error of Mean 1.512
Statistical Analysis 7: Comparison: Lapatinib + Trastuzumab + Aromatase Inhibitor (AI) vs Trastuzumab + Aromatase Inhibitor (AI); Physical well-being (PWB); Test type: Superiority; Least square difference = -1.46, 95% CI 2-sided [-2.82 to -0.11], Standard Error of Mean 0.690
Statistical Analysis 8: Comparison: Lapatinib + Aromatase Inhibitor (AI) vs Trastuzumab + Aromatase Inhibitor (AI); Physical well-being (PWB); Test type: Superiority; Least square difference = -1.54, 95% CI 2-sided [-2.90 to -0.18], Standard Error of Mean 0.693
Statistical Analysis 9: Comparison: Lapatinib + Trastuzumab + Aromatase Inhibitor (AI) vs Trastuzumab + Aromatase Inhibitor (AI); Social family wellbeing (SWB); Test type: Superiority; Least square difference = 0.39, 95% CI 2-sided [-1.01 to 1.79], Standard Error of Mean 0.711
Statistical Analysis 10: Comparison: Lapatinib + Aromatase Inhibitor (AI) vs Trastuzumab + Aromatase Inhibitor (AI); Social family wellbeing (SWB); Test type: Superiority; Least square difference = -0.55, 95% CI 2-sided [-1.96 to 0.86], Standard Error of Mean 0.715
Statistical Analysis 11: Comparison: Lapatinib + Trastuzumab + Aromatase Inhibitor (AI) vs Trastuzumab + Aromatase Inhibitor (AI); Emotional wellbeing (EWB); Test type: Superiority; Least square difference = 0.54, 95% CI 2-sided [-0.57 to 1.66], Standard Error of Mean 0.568
Statistical Analysis 12: Comparison: Lapatinib + Aromatase Inhibitor (AI) vs Trastuzumab + Aromatase Inhibitor (AI); Emotional wellbeing (EWB); Test type: Superiority; Least square difference = 0.40, 95% CI 2-sided [-0.72 to 1.53], Standard Error of Mean 0.571
Statistical Analysis 13: Comparison: Lapatinib + Trastuzumab + Aromatase Inhibitor (AI) vs Trastuzumab + Aromatase Inhibitor (AI); Functional wellbeing (FWB); Test type: Superiority; Least square difference = -0.99, 95% CI 2-sided [-2.26 to 0.28], Standard Error of Mean 0.646
Statistical Analysis 14: Comparison: Lapatinib + Aromatase Inhibitor (AI) vs Trastuzumab + Aromatase Inhibitor (AI); Functional wellbeing (FWB); Test type: Superiority; Least square difference = -1.32, 95% CI 2-sided [-2.60 to -0.04], Standard Error of Mean 0.649
Statistical Analysis 15: Comparison: Lapatinib + Trastuzumab + Aromatase Inhibitor (AI) vs Trastuzumab + Aromatase Inhibitor (AI); Breast cancer subscale (BCS); Test type: Superiority; Least square difference = -0.35, 95% CI 2-sided [-1.66 to 0.95], Standard Error of Mean 0.665
Statistical Analysis 16: Comparison: Lapatinib + Aromatase Inhibitor (AI) vs Trastuzumab + Aromatase Inhibitor (AI); Breast cancer subscale (BCS); Test type: Superiority; Least square difference = -0.83, 95% CI 2-sided [-2.14 to 0.48], Standard Error of Mean 0.668

10. Post Hoc Outcome: All Collected Deaths
Description: Pre-treatment deaths were collected from day of participant's informed consent to the day before first dose of study medication.
  On-treatment deaths were collected from first dose of study medication to 30 days after last dose of study medication (on-treatment), up to approximately 131 months.
  Deaths were collected in the post treatment survival follow up from 31 days after last dose of study medication until the end of the study, up to approximately 132 months.
Time Frame: Pre-treatment deaths: Up to 28 days prior to treatment. On-treatment deaths: Up to 131 months. Post-treatment deaths: up to 132 months.
Population: Intent-to-Treat (ITT) Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Lapatinib + Trastuzumab + Aromatase Inhibitor (AI) | Lapatinib + Aromatase Inhibitor (AI) | Trastuzumab + Aromatase Inhibitor (AI)
Number analyzed (Participants) | 124 | 123 | 122
Participants
  Pre-treatment deaths | 0 | 0 | 0
  On-treatment deaths: number analyzed (Participants) | 123 | 123 | 121
  On-treatment deaths | 5 | 8 | 5
  Post-treatment deaths: number analyzed (Participants) | 118 | 114 | 116
  Post-treatment deaths | 33 | 37 | 34
  All deaths | 38 | 45 | 39

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from first dose of study medication until the last dose plus 30 days post-treat follow-up, assessed up to approximately 131 months. Deaths were recorded from study start date until end of survival follow-up phase (end of study), assessed up to approximately 132 months.
Description: Deaths in the post-treatment survival follow-up were not considered adverse events. The total number at risk in the post-treatment survival included patients who entered this period. All-cause Mortality was assessed for all participants enrolled in the study, while Serious and Other Adverse Events were assessed for all participants who received at least one dose of the study medication.
Groups:
- Lapatinib + Trastuzumab + Aromatase Inhibitor (AI): Lapatinib + Trastuzumab + Aromatase Inhibitor (AI): Events up to 30 days post-treatment
- Lapatinib + Aromatase Inhibitor (AI): Lapatinib + Aromatase Inhibitor (AI): Events up to 30 days post-treatment
- Trastuzumab + Aromatase Inhibitor (AI): Trastuzumab + Aromatase Inhibitor (AI): Events up to 30 days post-treatment
- Lapatinib + Trastuzumab + Aromatase Inhibitor (AI) (Post-treatment): Lapatinib + Trastuzumab + Aromatase Inhibitor (AI) (Post-treatment): Deaths in the post-treatment survival follow-up were not considered adverse events
- Lapatinib + Aromatase Inhibitor (AI) (Post-treatment): Lapatinib + Aromatase Inhibitor (AI) (Post-treatment): Deaths in the post-treatment survival follow-up were not considered adverse events
- Trastuzumab + Aromatase Inhibitor (AI) (Post-treatment): Trastuzumab + Aromatase Inhibitor (AI) (Post-treatment): Deaths in the post-treatment survival follow-up were not considered adverse events
Arm/Group | Lapatinib + Trastuzumab + Aromatase Inhibitor (AI) | Lapatinib + Aromatase Inhibitor (AI) | Trastuzumab + Aromatase Inhibitor (AI) | Lapatinib + Trastuzumab + Aromatase Inhibitor (AI) (Post-treatment) | Lapatinib + Aromatase Inhibitor (AI) (Post-treatment) | Trastuzumab + Aromatase Inhibitor (AI) (Post-treatment)
All-Cause Mortality (participants affected / at risk) | 5/124 | 8/123 | 5/122 | 33/118 | 37/114 | 34/116
Serious Adverse Events (participants affected / at risk) | 27/123 | 23/123 | 14/121 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 113/123 | 107/123 | 86/121 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lapatinib + Trastuzumab + Aromatase Inhibitor (AI) (N=123) | Lapatinib + Aromatase Inhibitor (AI) (N=123) | Trastuzumab + Aromatase Inhibitor (AI) (N=121) | Lapatinib + Trastuzumab + Aromatase Inhibitor (AI) (Post-treatment) (N=0) | Lapatinib + Aromatase Inhibitor (AI) (Post-treatment) (N=0) | Trastuzumab + Aromatase Inhibitor (AI) (Post-treatment) (N=0)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | NA | NA | NA
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | NA | NA | NA
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | NA | NA | NA
Cardiac failure (Cardiac disorders) | 1 | 0 | 1 | NA | NA | NA
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 1 | NA | NA | NA
Cardiogenic shock (Cardiac disorders) | 0 | 1 | 0 | NA | NA | NA
Left ventricular dysfunction (Cardiac disorders) | 1 | 0 | 0 | NA | NA | NA
Anal fissure (Gastrointestinal disorders) | 0 | 1 | 0 | NA | NA | NA
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | NA | NA | NA
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | NA | NA | NA
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Asthenia (General disorders) | 0 | 0 | 1 | NA | NA | NA
Organ failure (General disorders) | 0 | 1 | 0 | NA | NA | NA
Pain (General disorders) | 1 | 0 | 0 | NA | NA | NA
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0 | NA | NA | NA
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0 | NA | NA | NA
Iodine allergy (Immune system disorders) | 1 | 0 | 0 | NA | NA | NA
Appendicitis (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Cellulitis (Infections and infestations) | 3 | 1 | 2 | NA | NA | NA
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | NA | NA | NA
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Osteomyelitis (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Pneumonia (Infections and infestations) | 0 | 1 | 0 | NA | NA | NA
Pyuria (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Sepsis (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Urinary tract infection (Infections and infestations) | 2 | 0 | 1 | NA | NA | NA
Urosepsis (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | NA | NA | NA
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | NA | NA | NA
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | NA | NA | NA
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | NA | NA | NA
Post procedural inflammation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | NA | NA | NA
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | NA | NA | NA
Alanine aminotransferase increased (Investigations) | 1 | 1 | 0 | NA | NA | NA
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | NA | NA | NA
Ejection fraction decreased (Investigations) | 7 | 1 | 2 | NA | NA | NA
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | NA | NA | NA
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | NA | NA | NA
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 | 0 | 0 | NA | NA | NA
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | NA | NA | NA
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | NA | NA | NA
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | NA | NA | NA
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | NA | NA | NA
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | NA | NA | NA
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | NA | NA | NA
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | NA | NA | NA
Ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | NA | NA | NA
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | NA | NA | NA
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | NA | NA | NA
Cognitive disorder (Nervous system disorders) | 0 | 1 | 0 | NA | NA | NA
Headache (Nervous system disorders) | 0 | 1 | 0 | NA | NA | NA
Intracranial aneurysm (Nervous system disorders) | 0 | 1 | 0 | NA | NA | NA
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | NA | NA | NA
Speech disorder (Nervous system disorders) | 0 | 0 | 1 | NA | NA | NA
Syncope (Nervous system disorders) | 1 | 0 | 0 | NA | NA | NA
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | NA | NA | NA
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | NA | NA | NA
Pyelocaliectasis (Renal and urinary disorders) | 1 | 0 | 0 | NA | NA | NA
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | NA | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | NA | NA | NA
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | NA | NA | NA
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | NA | NA | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | NA | NA | NA
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | NA | NA | NA
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | NA | NA | NA
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | NA | NA | NA
Thrombophlebitis (Vascular disorders) | 0 | 1 | 0 | NA | NA | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lapatinib + Trastuzumab + Aromatase Inhibitor (AI) (N=123) | Lapatinib + Aromatase Inhibitor (AI) (N=123) | Trastuzumab + Aromatase Inhibitor (AI) (N=121) | Lapatinib + Trastuzumab + Aromatase Inhibitor (AI) (Post-treatment) (N=0) | Lapatinib + Aromatase Inhibitor (AI) (Post-treatment) (N=0) | Trastuzumab + Aromatase Inhibitor (AI) (Post-treatment) (N=0)
Anaemia (Blood and lymphatic system disorders) | 8 | 7 | 8 | NA | NA | NA
Neutropenia (Blood and lymphatic system disorders) | 6 | 7 | 3 | NA | NA | NA
Abdominal pain upper (Gastrointestinal disorders) | 9 | 7 | 9 | NA | NA | NA
Cheilitis (Gastrointestinal disorders) | 7 | 1 | 0 | NA | NA | NA
Diarrhoea (Gastrointestinal disorders) | 87 | 64 | 11 | NA | NA | NA
Dyspepsia (Gastrointestinal disorders) | 8 | 4 | 0 | NA | NA | NA
Nausea (Gastrointestinal disorders) | 28 | 28 | 13 | NA | NA | NA
Stomatitis (Gastrointestinal disorders) | 23 | 16 | 5 | NA | NA | NA
Vomiting (Gastrointestinal disorders) | 16 | 19 | 1 | NA | NA | NA
Asthenia (General disorders) | 15 | 7 | 6 | NA | NA | NA
Fatigue (General disorders) | 15 | 19 | 12 | NA | NA | NA
Oedema peripheral (General disorders) | 8 | 5 | 5 | NA | NA | NA
Pyrexia (General disorders) | 7 | 6 | 6 | NA | NA | NA
Nasopharyngitis (Infections and infestations) | 8 | 6 | 10 | NA | NA | NA
Paronychia (Infections and infestations) | 39 | 21 | 0 | NA | NA | NA
Upper respiratory tract infection (Infections and infestations) | 13 | 8 | 7 | NA | NA | NA
Urinary tract infection (Infections and infestations) | 7 | 0 | 5 | NA | NA | NA
Alanine aminotransferase increased (Investigations) | 11 | 20 | 9 | NA | NA | NA
Aspartate aminotransferase increased (Investigations) | 11 | 22 | 11 | NA | NA | NA
Blood alkaline phosphatase increased (Investigations) | 5 | 7 | 9 | NA | NA | NA
Blood bilirubin increased (Investigations) | 3 | 8 | 1 | NA | NA | NA
Ejection fraction decreased (Investigations) | 10 | 3 | 3 | NA | NA | NA
Weight decreased (Investigations) | 12 | 13 | 3 | NA | NA | NA
Decreased appetite (Metabolism and nutrition disorders) | 22 | 18 | 4 | NA | NA | NA
Hypokalaemia (Metabolism and nutrition disorders) | 9 | 8 | 0 | NA | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 22 | 19 | 15 | NA | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 12 | 10 | NA | NA | NA
Bone pain (Musculoskeletal and connective tissue disorders) | 7 | 4 | 7 | NA | NA | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 6 | 8 | NA | NA | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 | 12 | 5 | NA | NA | NA
Dizziness (Nervous system disorders) | 10 | 10 | 9 | NA | NA | NA
Headache (Nervous system disorders) | 9 | 21 | 15 | NA | NA | NA
Insomnia (Psychiatric disorders) | 5 | 12 | 4 | NA | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 16 | 17 | NA | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 9 | 8 | NA | NA | NA
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10 | 8 | 0 | NA | NA | NA
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 7 | 3 | 1 | NA | NA | NA
Alopecia (Skin and subcutaneous tissue disorders) | 14 | 8 | 2 | NA | NA | NA
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 16 | 11 | 2 | NA | NA | NA
Dry skin (Skin and subcutaneous tissue disorders) | 11 | 11 | 0 | NA | NA | NA
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 13 | 11 | 1 | NA | NA | NA
Pruritus (Skin and subcutaneous tissue disorders) | 11 | 11 | 2 | NA | NA | NA
Rash (Skin and subcutaneous tissue disorders) | 43 | 36 | 3 | NA | NA | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7 | 7 | 0 | NA | NA | NA
Skin fissures (Skin and subcutaneous tissue disorders) | 7 | 3 | 2 | NA | NA | NA
Hypertension (Vascular disorders) | 9 | 4 | 8 | NA | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.